CLINICAL TRIAL: NCT05022381
Title: Radiofrequency Thermocoagulation to the Articular Branches of the Femoral and Obturatory Nerve in Chronic Hip Pain
Brief Title: Treatment of Chronic Hip Pain by Application of Conventional Radiofrequency Thermocoagulation to the Articular Branches of the Femoral and Obturatory Nerve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, sevilay şimşek, Resident doctor, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/04
Record Dates: First submitted 2021-08-25; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hip Pain Chronic
Keywords: chronic hip pain; Radiofrequency thermocoagulation; Algology; femoral and obturatuar nerve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative and Postoperative Pain Level (Other): The preoperative pain level, hip function and quality of life of patients who underwent radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerve in chronic hip pain will be compared with the postoperative pain level, hip function and quality of life of these patients.
  Interventions: Procedure: Radiofrequency thermal coagulation of articular branches of femoral and obturator nerves

INTERVENTIONS:
Procedure: Radiofrequency thermal coagulation of articular branches of femoral and obturator nerves — Patients are operated under sedation in the operating room. C-arm fluoroscopy device is used for imaging purposes for radiofrequency thermocoagulation process. In order to prevent vascular injury, the needle is advanced under the guidance of ultrasonography. There are target points determined in fluoroscopy for the femoral nerve and the obturatory nerve. Before the thermocoagulation procedure, local anesthetic and steroid are injected into each of the target points. Patients who do not have any complications after the procedure and who are mobilized are discharged in the 2nd hour.

SUMMARY:
The estimated prevalence of hip joint pain is 7% in men and 10% in women over the age of 45 years.Although physical therapy and weight loss, use of walking aids (such as walking sticks) and analgesic agents are used as conservative treatment methods, these methods usually provide short-term and partial benefits.The anterior sensory innervation of the hip joint is provided by the articular branches of the femoral and obturatory nerve. Denervation of the articular branches of the femoral and obturator nerves with the radiofrequency thermocoagulation (RFT) method is a method used in chronic hip pain. In this study, we aimed to show the decrease in pain levels and the effect on quality of life of patients who underwent hip RFT.

DETAILED DESCRIPTION:
Hip pain is a common medical condition with increasing age.The effectiveness of conservative methods used in hip pain is limited.Since the lifespan of prostheses used in hip surgery is limited, new methods are needed in the treatment of pain.The anterior sensory innervation of the hip joint is provided by the articular branches of the femoral and obturatory nerve. Denervation of the articular branches of the femoral and obturator nerves with the radiofrequency thermocoagulation (RFT) method is a method used in chronic hip pain.In previous studies with small groups, it was shown that radiofrequency thermocoagulation procedure caused 50% reduction in hip pain between 1-11 months.Hip joint radiofrequency thermocoagulation is a procedure applied in our clinic. In this study, we aimed to show the decrease in pain levels and the effect on quality of life of patients who underwent hip RFT.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. Written consent has been obtained
3. Those with chronic hip pain for more than 3 weeks

Exclusion Criteria:

1. Major psychiatric illness
2. The patient has lumbar compression pain or referred pain
3. Patients using anticoagulant agents
4. Patients with infection in the area to be treated
5. Those who are allergic to local anesthetics
6. Those who are allergic to betamethasone
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Chronic pain level | 1 month,3 month, 6 month
  For this, the patients' preoperative, 1st month, 3rd month and 6th month VPS (Verbal Pain Score) scores will be checked. A 50% reduction in the verbal pain score will be considered significant.

SECONDARY OUTCOMES:
Hip functional capacity | 1month,3 month,6month
  For this purpose, the WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale will be checked at the 1st, 3rd, 6th, 6th months in order to evaluate the functional capacity before the procedure.

OTHER OUTCOMES:
Life Quality | 1month, 3 month,6 month
  For this purpose, patients will be subjected to the Short Form-12- test, which is a short scale of quality of life at 1st month, 3rd month and 6th month.
Acute pain | 1 week
  Week 1 Verbal Pain Score will be checked to observe the improvement in acute pain in patients. A 50% decrease in verbal pain score will be considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No